CLINICAL TRIAL: NCT07294378
Title: Evaluation of the Dental Changes Associated With the Traction of Palatally Impacted Canines Using the Conventional Versus the Corticotomy-assisted Method: A Randomized Controlled Trial
Brief Title: Dental Changes Following the Traction of Impacted Maxillary Canines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-2025-Ortho-11
Record Dates: First submitted 2025-12-07; First posted 2025-12-19 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Impaction of Tooth
MeSH Terms: conditions — Tooth, Impacted | interventions — Piezosurgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Accelerated canine traction group (Experimental): Perforations of the bone surrounding the impacted canine will be conducted at the time of canine exposure. Two months later, another flapless corticotomy procedure will be performed during the withdrawal of the impacted canine.
  Interventions: Procedure: Corticotomy
- Conventional canine traction (Active Comparator): The canines will be withdrawn to the dental arch using the conventionnal method without subjecitng the patient to any additional surgical intervention.
  Interventions: Procedure: Conventional traction

INTERVENTIONS:
Procedure: Corticotomy — During the surgical exposure phase in the acceleration group, the cortical bone will be perforated around the exposed canine crown (6-8 holes) wherever possible-this procedure aims to accelerate the withdrawal movement of the impacted canine. A 1 mm round bur will be used to create circular holes (1 mm in diameter, 1-2 mm in depth, and spaced about 1.5 mm apart). After two months of the surgical exposure, the second acceleration procedure will be performed. Two or three vertical incisions (8 mm height) will be made using a surgical scalpel at the buccal side of the impaction area. The cortical cuts (2-3 mm in depth, 1 mm in width, and spaced about 2 mm apart) will be performed using a flapless piezosurgery technique along the vertical lines.
  Other Names: flapless corticotomy; piezocision; piezosurgery
  Arms: Accelerated canine traction group
Procedure: Conventional traction — The canines will be withdrawn using conventional methods without any surgical acceleration.
  Arms: Conventional canine traction

SUMMARY:
The impaction of maxillary canines is a challenge for orthodontists. Recently, new methods have been proposed to accelerate canine withdrawal. The associated dental changes between the conventional and accelerated methods of canine traction have not yet been assessed.

DETAILED DESCRIPTION:
Impacted canines are defined as those that have not erupted within 6 six months after completing the formation of their roots or that were not present within the dental arch during their eruption phase. Upper Impacted canines are present in 2% of the general population and occur in females at a rate of 1.17%, which is almost twice the incidence in males. The incidence of palatal impaction ranges from 60% to 80% and is present bilaterally with a rate of 75-95%. The upper canines usually erupt at an average age of 10.5 years in females and 11.5 years in males, with an individual difference of 3-4 years. Eruption failure of the upper canines occurs because of hard or soft tissue obstructions or an abnormal eruption pathway.

The most important causes of palatally impaction of upper canines are dental arch length deficiency, over-retained primary teeth, and trauma during the canine formation stage. One local mechanical cause is a decrease in the width of the upper dental arch. McConnell et al. reported that patients with upper impacted canines had a reduction in dental arch width, especially in the anterior region. On the other hand, unilateral or bilateral upper canine impaction can affect upper dental arch width and alter smile symmetry.

The impaction of the upper canine is also considered as one of the causes that lead to a lack of transverse development of the maxillary dental arch, especially the inter-premolar width. This is supported by the functional matrix theory, which considers that the presence of the organ stimulates bone growth. Thus, the natural eruption of the canine stimulates the normal transverse growth of the dental arch.

Many treatment strategies were used to treat impacted canine cases, but orthodontic traction after surgical exposure was the most commonly recommended method in the literature, given the great aesthetic and functional value of the upper canines. Two main surgical methods are used for this purpose: the open and closed surgical approaches.

Several mechanical means have been used to obtain the traction force. However, choosing the appropriate mechanical method that produces the least undesirable effects on adjacent teeth was a challenge for the clinical practitioner.

Many factors could result in unwanted changes in the spatial position of the adjacent teeth, such as the use of an open coil spring, direct reliance on these teeth to tract the impacted canine, the type of baseline orthodontic archwire used, and the type of orthodontic anchorage means. These side effects on adjacent teeth can be minimized by using techniques such as the segmented archwire technique and temporary anchorage devices (TADs).

ELIGIBILITY:
Inclusion Criteria:

1. patients' ages ranged from 18 to 28 years old
2. unilaterally palatally or mid-alveolar upper impacted canine
3. patients who have never received orthodontic treatment previously
4. mild crowding of the maxillary arch (less than 4 mm) and class I first molars relation

Exclusion Criteria:

1. bilateral or buccal canine impaction
2. patients who have a contraindication to perform oral surgery under local anesthesia (social, psychological, mor edical)
3. more than 45-degree angle between the longitudinal axis of the impacted canines and the facial midline
4. bad oral health

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2023-03-02 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2025-01-19 (Actual)

PRIMARY OUTCOMES:
Change in the upper dental midline deviation | T1: before the commencement of canine traction (expected to occur within 3-5 months following the beginning of fixed orthodontic treatment). T2: at the end of the canine traction stage (expected to occur with 5-8 months after T1)
  The deviation of the upper dental midline will be measured in millimeters as the distance from the maxillary central incisors contact point to the maxillary model midline. This will be performed on the plaster models.
Change in the rotation of the lateral incisor. | T1: before the commencement of canine traction (expected to occur within 3-5 months following the beginning of fixed orthodontic treatment). T2: at the end of the canine traction stage (expected to occur with 5-8 months after T1)
  The rotation will be measured in degrees as the angle between the maxillary model midline and the line connecting the mesial-distal marginal points of the adjacent lateral incisor.
Change in the rotation of the first premolar | T1: before the commencement of canine traction (expected to occur within 3-5 months following the beginning of fixed orthodontic treatment). T2: at the end of the canine traction stage (expected to occur with 5-8 months after T1)
  The rotation will be measured in degrees as the angle between the maxillary model midline and the line connecting the mesial-distal marginal points of the adjacent first premolar.
Change in the inter-premolar width | T1: before the commencement of canine traction (expected to occur within 3-5 months following the beginning of fixed orthodontic treatment). T2: at the end of the canine traction stage (expected to occur with 5-8 months after T1)
  Inter-premolar width will be measured in millimeters as the distance from the deepest point in the central groove of the adjacent first premolar and its counterpart on the contralateral side

CONTACTS AND LOCATIONS:
Overall Officials: Mahran Raheel Mousa, DDS, MSc, PhD, Principal Investigator — Department of Orthodontics, Faculty of Dentistry, Al-Hawash Private University, Homs, Syria; Mohammad Younis Hajeer, DDS, MSc, PhD, Study Director — Department of Orthodontics, Faculty of Dentistry, Damascus University; Omar Ahmad Heshmeh, DDS, MSc, PhD, Study Director — Department of Oral and Maxillofacial Surgery, Faculty of Dentistry, Damascus University
Locations (1):
- Orthodontics Department, Faculty of Dentistry, Damascus, Rif-dimashq Governorate, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fischer TJ. Orthodontic treatment acceleration with corticotomy-assisted exposure of palatally impacted canines. Angle Orthod. 2007 May;77(3):417-20. doi: 10.2319/0003-3219(2007)077[0417:OTAWCE]2.0.CO;2. PMID 17465647
- [Background] Alyafrusee ES, Zheng B, Almashraqi AA, Almaqrami BS, Yang X, Xu H, Alhammadi MS, Liu Y. Three-dimensional dentoalveolar characteristics of a labially impacted dilacerated maxillary central incisor using cone-beam computed tomography. Sci Rep. 2025 Jul 9;15(1):24669. doi: 10.1038/s41598-025-10043-9. PMID 40634539
- [Background] Hocevar M, Ovsenik M, Golez A. Position of Maxillary Lateral Incisor and First Premolar in Impaction of Maxillary Canines: A Controlled Clinical CBCT and 3D Study Model Analysis. Dent J (Basel). 2025 Oct 27;13(11):497. doi: 10.3390/dj13110497. PMID 41294478
- [Background] Mousa MR, Hajeer MY, Burhan AS, Heshmeh O. Adult periodontal comparison after treatment of palatally impacted canines aligned by conventional or accelerated minimally-invasive corticotomy-assisted orthodontic traction: A randomized controlled trial. Int Orthod. 2023 Sep;21(3):100785. doi: 10.1016/j.ortho.2023.100785. Epub 2023 Jun 15. PMID 37329591
- [Background] Mousa MR, Hajeer MY, Burhan AS, Heshmeh O, Alam MK. The effectiveness of minimally-invasive corticotomy-assisted orthodontic treatment of palatally impacted canines compared to the traditional traction method in terms of treatment duration, velocity of traction movement and the associated dentoalveolar changes: A randomized controlled trial. F1000Res. 2023 Jun 19;12:699. doi: 10.12688/f1000research.135338.1. eCollection 2023. PMID 37920456